CLINICAL TRIAL: NCT00296868
Title: Prophylactic Administration of Vitamin C in Wrist Fractures; a Randomized Placebo Controlled Multicentre Dose-Finding Study of the Incidence of Complex Regional Pain Syndrome
Brief Title: Prophylactic Administration of Vitamin C in Wrist Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stichting Achmea Slachtoffer en Samenleving (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SRvB/2001-290/JV
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2006-02-27 (Estimated); Status verified 2005-12

CONDITIONS: RSD (Reflex Sympathetic Dystrophy); Algodystrophy; CRPS Type I
Keywords: reflex sympathetic dystrophy; ascorbic acid; primary prevention; radius fractures
MeSH Terms: conditions — Complex Regional Pain Syndromes; Reflex Sympathetic Dystrophy; Radius Fractures | interventions — Ascorbic Acid

INTERVENTIONS:
Drug: ascorbic acid (vitamin C) versus placebo

SUMMARY:
Complex Regional Pain Syndrome or posttraumatic dystrophy is a pain syndrome which develops after a trauma, surgery or for unknown reason. The incidence after wrist fractures varies in literature from 2 - 37%. The female sex is involved three times as much as the male sex. There is one study in literature which describes a prophylactic effect of vitamin C after wrist fractures. Goal of this study is to search for a dose dependent effect of vitamin C and to replicate these earlier findings.

DETAILED DESCRIPTION:
The trial was designed as a multicentre, randomized, controlled study. Three hospitals in the Netherlands participated in this study, using the same experimental design.

Adults (18 years or above) with a wrist fracture who were seen in the emergency department of each hospital were asked to participate in this study. Patients were asked to start the trial medication on the day of the fracture. Two capsules had to be taken once daily for 50 days. Patients were allocated randomly to receive either placebo or a dosage of 200, 500 or 1500 mg of vitamin C daily.

The endpoint of the study was defined as the presence of CRPS at any moment, in the period up to one year after the fracture. All participants and physicians were unaware of the treatment allocation.

Patients were seen after 1 week, 4 or 5 weeks (or when the cast was removed), 6 or 7 weeks, 12 weeks, and 26 weeks. After one year patients were interviewed by telephone or received an inquiry letter with a postage-paid envelope for their reply. The normal fracture treatment, either conservative or operative, was not compromised by the protocol, and if necessary patients were seen more often and/or at other times than planned.

Complex regional pain syndrome was diagnosed when four of the following five symptoms were present throughout an area larger than the wrist, including the area distal to the wrist (hand and fingers), and if they occurred or increased after activity: unexplained diffuse pain, which is not in normal relation to the fracture; difference in skin color relative to the other arm; diffuse edema; difference in skin temperature relative to the other arm; limited active range of motion, unrelated to the stage of fracture treatment. If CRPS was diagnosed, the end point of the study was reached and the protocol was terminated to enable treatment for CRPS.

ELIGIBILITY:
Inclusion Criteria:

* wrist fracture
* adult (18 years and older)

Exclusion Criteria:

* no comprehension of the written information
* not able to appear for follow-up (living abroad)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-01; Study Completion 2005-12

PRIMARY OUTCOMES:
the existence of CRPS until one year after follow-up

SECONDARY OUTCOMES:
difference in outcome and dose (dose comparison) after one year of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Zollinger, MD, Principal Investigator — department of orthopedic surgery, Ziekenhuis Rivierenland, Pres Kennedylaan 1, 4002 WP Tiel, the Netherlands
Locations (1):
- Rode Kruis Ziekenhuis, Vondellaan 13, Beverwijk, Netherlands

REFERENCES:
- [Result] Zollinger PE, Tuinebreijer WE, Kreis RW, Breederveld RS. Effect of vitamin C on frequency of reflex sympathetic dystrophy in wrist fractures: a randomised trial. Lancet. 1999 Dec 11;354(9195):2025-8. doi: 10.1016/S0140-6736(99)03059-7. PMID 10636366